CLINICAL TRIAL: NCT05705258
Title: Special Drug Use Investigation for Eylea for Retinopathy of Prematurity (ROP)
Brief Title: A Study to Collect Data on the Use of Eylea in Babies Born Too Early Who Have a Condition of the Eye Where Blood Vessels Grow Abnormally in the Retina (Retinopathy of Prematurity)
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22069
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Retinopathy of Prematurity; Newborns; Infants
Keywords: ROP
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept treatment: The patients will be included in this study by investigators who are prescribing Aflibercept (AFL) routinely in their clinical practice. The enrollment of each patient in this study is able to accept at latest in 6 months from initiation of treatment.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Treatment with Intravitreal (IVT)-AFL must be made by the treating ophthalmologist

SUMMARY:
This is an observational study to collect data from Japanese babies with retinopathy of prematurity (ROP) who will be treated with Eylea. In observational studies, only observations are made without specified advice or interventions.

ROP is a condition that affects the eye and occurs only in babies who are born too early. Most cases of ROP are mild and get better without treatment, but more serious cases need to be treated in time. ROP happens when the blood vessels in the "retina" grow abnormally. The retina is the layer of tissue at the back of the eye that picks up light and sends messages to the brain. In babies with ROP, these abnormal blood vessels can leak. This causes damage to the retina and can sometimes move it out of place causing medical problems such as blindness.

Eylea is received as an injection into the eye. It works by blocking a certain protein (VEGF) that can cause blood vessels in the retina to grow abnormally. Eylea is already available in Japan and is approved for doctors to prescribe to babies with ROP.

The participants in this study are Japanese babies with ROP that their doctors decided to treat with Eylea before the start of this study. Babies with ROP that were already prescribed Eylea by their doctors may also be included.

The main purpose of this study is to collect more data on how safe the treatment with Eylea is in babies with ROP under a real-world setting. Another purpose of this study is to collect more data on how well Eylea works in these participants.

To see how safe Eylea is, the study doctors will collect all medical problems that the participants treated with Eylea have. These medical problems are called adverse events. Doctors keep track of all the adverse events that happen, even if they do not think that they might be related to the treatment.

To see how well Eylea works, the study doctors will check the number of participants:

* with no active ROP after starting treatment
* where ROP came back up to 6 months after start of treatment

In this study, the study doctor will:

* collect past data of the participants from medical records
* interview the participants
* collect treatment-related data during routine visits. The study duration is 6 months with 3 planned visits. One visit will be at start of treatment, one at one month and one at 6 months after start of treatment. All data required for this study will be collected during routine visits. Besides this data collection, no further tests or examinations are planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ROP requiring treatment
* Patients who have received IVT-AFL treatment according to Japanese approved labeling for AFL in ROP.
* ICF obtained from legal representative.

Exclusion Criteria:

* Patients who have contradictions based on approved label
* Patients who have received IVT-AFL treatment before the treatment for the enrollment Patient.
* Diagnosis of other indication

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a diagnosis of ROP will be enrolled after the decision for treatment with AFL has been made by the investigator.
  Patients who have been prescribed AFL in accordance with the product label in Japan will be eligible to be enrolled. Indications and contraindications according to the local market authorization should be carefully considered.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of any treatment-emergent adverse events (TEAEs) | Up to 6 months after initiation of Aflibercept

SECONDARY OUTCOMES:
Proportion of patients who improvement of the activity of ROP | At month 1 or month 6 after initiation of Aflibercept
  Active ROP will be assessed by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/